CLINICAL TRIAL: NCT05795790
Title: Observational Cross-sectional Study to Define the Role of Serology and Other Immunological Tests in the Diagnosis of COVID-19 in the Pediatric Population
Brief Title: Serology and Other Immunologic Response Tests in the Diagnosis of COVID-19 in Pediatrics
Acronym: Covid_IMMUNO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Other Study IDs: RC 35/20
Record Dates: First submitted 2023-03-28; First posted 2023-04-03 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: COVID-19
Keywords: COVID-19; Pediatrics; Immunology
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: None Retained — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Despite the SARS-CoV-2 virus being present worldwide, and although it is now clear that children are affected by the disease with milder symptoms than adults, many immunological questions, which are very relevant for Public Health reasons and for the organization of services, remain unsolved. The role of serology for the diagnosis of COVID-19, particularly in the pediatric age, is still very uncertain. Preliminary evidence suggests that not all children with SARS-Cov-2 infection develop antibody levels that can be detected by currently employed methods. This makes it crucial to identify other methodologies that are able to evaluate the true prevalence of prior SARS-CoV-2 infection in the pediatric population. Many other aspects of the immunological mechanisms of response to SARS-CoV-2 are also uncertain, such as the role of cellular immunity, and generally the role of immunity (cellular and antibody) in protecting against the disease in the medium and long term. Finally, questions remain open regarding cross-immunity with other previously circulating coronaviruses and their impact on the pediatric population in terms of protection against COVID-19 infection, disease development, or reinfection. This study aims to help clarify the role of serology and other immune response tests in the diagnosis of COVID-19 in the pediatric population. Specifically, it aims to assess: the prevalence of SARS-CoV-2 seroconversion cases among the pediatric population accessing the National Health System (NHS), at different moments in time and in different regions of Italy; whether cellular immunity tests can help to identify children who have had SARS-CoV-2 infection, particularly children with low antibody levels, and thus to better estimate the prevalence of prior SARS-CoV-2 infection; the prevalence of cross-reactivity with other coronaviruses; whether immunity (antibody and cellular) is protective in the medium/long term; and if there are healthy carriers, i.e. individuals who have had prior SARS-CoV-2 infection, who are asymptomatic but may harbor SARS-CoV-2 in the pharynx, with the risk of transmitting it.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-17 years
* Access to National Health System facilities for blood collection.

Exclusion Criteria:

* Immunodepression (primary or secondary)
* Refusal to participate in the study

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Pediatric subjects (0-17 years) accessing National Health System facilities for blood collection
Sampling Method: Non-Probability Sample
Enrollment: 249 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of SARS-CoV-2 seroconversion | Through study completion, an average of 3 years
  In blood samples collected among the pediatric population accessing the National Health System at different times and in different regions of Italy

SECONDARY OUTCOMES:
Prevalence of subjects with a cellular T response to SARS-CoV-2 | Through study completion, an average of 3 years
  In blood samples collected among the pediatric population accessing the National Health System at different times and in different regions of Italy
Prevalence of cross-reactivity with other coronaviruses | Through study completion, an average of 3 years
  In blood samples collected among the pediatric population accessing the National Health System at different times and in different regions of Italy
Frequency of activation of IgG-type immunity (antibody and cellular) in children testing positive for SARS-CoV-2 at nasopharyngeal swab | Through study completion, an average of 3 years
  In blood samples collected among the pediatric population accessing the National Health System at different times and in different regions of Italy
Persistence of positivity for SARS-CoV-2 at nasopharyngeal swab | Through study completion, an average of 3 years
  Among the pediatric population accessing the National Health System at different times and in different regions of Italy

CONTACTS AND LOCATIONS:
Overall Officials: Marzia Lazzerini, MD, Study Director — IRCCS materno infantile Burlo Garofolo
Locations (1):
- IRCCS Burlo Garofolo, Trieste, Italy